CLINICAL TRIAL: NCT02845050
Title: Phase Ib/II Study Assessing the Neo-adjuvant Combination Therapy of Vinflunine With Cisplatin Followed by Radical Cystectomy in Patients With Muscle-invasive Bladder Cancer (JaNEO)
Acronym: JaNEO
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participants found
Sponsor: Ligartis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JaNEO-001; 2016-000081-33 (EudraCT Number)
Record Dates: First submitted 2016-07-12; First posted 2016-07-27 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Bladder Cancer
Keywords: neo-adjuvant; vinflunine; cisplatin; radical cystectomy; muscle-invasive bladder cancer; JaNEO
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — vinflunine; Cisplatin; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinflunine+Cisplatin+radical cystectomy (Experimental): neoadjuvant combination of Vinflunine+Cisplatin before radical cystectomy as proof of principle (one arm only!)
  Interventions: Drug: Vinflunine; Drug: Cisplatin; Procedure: Radical cystectomy

INTERVENTIONS:
Drug: Vinflunine — One cycle is defined as a period of 3 weeks of treatment:
  Vinflunine (280 mg/m²) on Day 1, every 21 days as a 20 minute IV infusion
  Cisplatin (70 mg/m²) on Day 2, every 21 days
  4 cycles of neo-adjuvant chemotherapy prior to radical cystectomy
Drug: Cisplatin — One cycle is defined as a period of 3 weeks of treatment:
  Vinflunine (280 mg/m²) on Day 1, every 21 days as a 20 minute IV infusion
  Cisplatin (70 mg/m²) on Day 2, every 21 days
  4 cycles of neo-adjuvant chemotherapy prior to radical cystectomy
Procedure: Radical cystectomy — max. 4 weeks after 4 cycles of neo-adjuvant treatment radical cystectomy will be performed

SUMMARY:
Phase Ib/II study assessing the neo-adjuvant combination therapy of vinflunine with cisplatin followed by radical cystectomy in patients with muscle-invasive bladder cancer (JaNEO).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years and ≤ 75 years with legal capacity
2. Signed written informed consent
3. Histologically confirmed muscle-invasive urothelial cell carcinoma of the bladder (MIBC) with clinical T2-T4a (N0/Nx, M0) assessed by primary PDD-guided TUR-B and by the screening imaging (MRI pelvis and CT chest/abdomen) which both must include the use of contrast medium
4. Confirmed adequate complete resection of all visible tumor during TUR-B according to current treatment guidelines before registration; the latest TUR-B must have been done ≤ 8 weeks before registration
5. ECOG performance status of 0 or 1
6. Adequate bone marrow, renal and hepatic functions as evidenced by the following:

   * Absolute Neutrophil Count ≥ 2,000 mm3 and ≤ 7,500 mm3
   * Hemoglobin ≥ 12 g/dL for the safety phase of the study; if the study treatment proved to be adequate tolerated during this safety phase, the threshold can be lowered to ≥ 10 g/dL according to the decision of the study steering committee
   * Platelet count ≥ 100,000 mm3
   * Serum albumin within normal range
   * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Transaminases (ALT, AST) ≤ 1.5 x ULN
   * Creatinine clearance ≥ 60 mL/min, calculated based on a 24h-measured creatinine clearance
   * Serum Urea < 25 mg/100 ml
7. Absence of psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; these conditions should be assessed with the patient before registration
8. Electrocardiogram (ECG) without modifications that suggest a high risk of occurrence of an acute clinical event (such as signs of angina pectoris or high-risk arrhythmia, etc.); cardiologist consultation is required, if relevant abnormalities are observed in the screening ECG-assessment

Exclusion Criteria:

1. Prior systemic chemotherapy for any kind of malignancy; prior intravesical chemotherapy or treatment with BCG is allowed
2. Prior radiation of the pelvis or any prior radiation to ≥ 30 % of the bone marrow
3. Evidence of lymph node (N+) or distant metastasis (M1) in the screening imaging assessment, including known brain metastases or leptomeningeal involvement (however, brain-MRI-scans are not required to rule out CNS-involvement, unless there is clinical suspicion of central nervous system (CNS) disease)
4. Any contraindication with regard to contrasted imaging (MRI or CT)
5. Other malignancies except adequately treated basal carcinoma of the skin, localized prostate cancer Gleason ≤ 6, in-situ cervix carcinoma or any other tumor with a disease free interval ≥ 5 years
6. Peripheral neuropathy Grade ≥ 2 NCI CTCAE v4.03 or hearing impairment Grade ≥ 2 NCI CTCAE v.4.03
7. Any concurrent chronic system immune therapy or previous organ allograft
8. Weight loss > 5 % within the last 3 months before registration
9. Any other serious illness or medical condition including:

   * Infection requiring systemic anti-infective therapy within the last 2 weeks before registration
   * History of cardio-vascular disease that might compromise the safe administration of cisplatin
   * Dehydration requiring IV fluid substitution
   * Any medical condition that might not be controlled, e.g. patients with unstable angina pectoris, myocardial infarction < 6 months before registration or uncontrolled diabetes, congestive cardiac failure > NYHA grade I
10. Known hypersensitivity to the study drugs or to drugs with similar chemical structures
11. Treatment with any potent CYP3A4 inhibitor or inductor (e.g. ketoconazole, itraconazole, ritonavir, amprenavir, indinavir, rifampicine) or phenytoine; replacement of such treatment with alternative treatment options before start of study treatment is acceptable, if medically feasible and ethically acceptable
12. 12. Treatment with any medication that is known to prolong the QT/QTc interval and/or to cause Torsades de Pointes (e.g. azithromycine, amitryptiline, imipramine, clozapine, flu-ox¬etine, cisapride); replacement of such treatment with alter¬na¬ti¬ve options before start of study treatment is acceptable, if medically feasible and ethically acceptable
13. Treatment with hexamethylmelamin, pyridoxine, penicillamine or any other drug with known potential to affect the efficacy of cisplatin
14. Treatment with any other investigational or anti-cancer therapy ≤ 30 days before registration
15. Pregnant or lactating female patients or female patients of childbearing potential with positive pregnancy test at screening
16. Women of child-bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 6 months after the study
17. Sexually active fertile men, who are unwilling or unable to use an effective birth control from day of informed consent and for up to 6 months after the last cycle of chemotherapy, if their partners are women of child-bearing potential (if cystectomy is not performed) effective birth control means the use of condoms ideally combined with any acceptable contraception of the male patient's partner as described in exclusion criterion 16

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | cystectomy
  Rate of pathological complete response (pCR) at cystectomy assessed by central pathological review (Prof. Hartmann, Erlangen), if the initial safety phase allows continuation of the trial with the phase II part

SECONDARY OUTCOMES:
Overall radiological response rate before cystectomy | prior cystectomy
  RECIST v1.1
Progression rate | after 2 and 4 cycles (of 21 days length) of treatment
  RECIST v1.1
Safety of chemotherapy measured by adverse events and clavien-dindo grades | through study completion after 12 months-follow up
  An evaluation of adverse events and serious adverse events will be done. Alle analyses of adverse events will be done using the CTCAE-classification v4.03. Events of grade 3-4 will be evaluated seperatly. Also, all events reported to be related to cystectomy will be evaluated using the clavien-dindo-grades.
Rate of complications at cystectomy | at cystectomy
Perioperative morbidity/mortality | 30 days and 90 days post surgery
Cancer-specific survival | one year after cystectomy
  Evaluation will be done from date of study registration to death on disease or the last visit date (if not death at timepoint of evaluation). Patients that died due to other reasons than cancer will be evaluated with their last date known alive.
QoL - GIQLI | Cycle 1-4 Day 1+ cystectomy + 1,3 and 12 months after cystectomy
  If Values for total or subscale scores are missing, no imputation will be applied. To summarize scored scales descriptive statistics will be used. Patients with an evaluable baseline score and at least one evaluable post baseline score will be included into analyses to evaluate changes from baseline.
QoL - QLQ-C30 | Cycle 1-4 Day 1+ cystectomy + 1,3 and 12 months after cystectomy
  If Values for total or subscale scores are missing, no imputation will be applied. To summarize scored scales descriptive statistics will be used. Patients with an evaluable baseline score and at least one evaluable post baseline score will be included into analyses to evaluate changes from baseline.

OTHER OUTCOMES:
Relapse rate and location of relapse not RECIST-standardized | at 1 month, 3 months and 1 year after cystectomy
  Evaluated will be the number of patients with relapse 1, 3 and 12 months after cystectomy. The same evaluation will be done seperately for different locations of relapse, e. g. local relapse, distant metastases (lung, liver, bone, extraregional lymp nodes)
Biobanking | Day 1 of cyle 1-4, Day 15 of cyle 1, at cystectomy, 1, 3 and 12 months follow up, and baseline for tumour tissue
  Blood, urine and tissue will be collected in a biobank for further evaluations that are not determined yet.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Dept. Urology, University Hospital Marburg, Marburg/ Lahn, Baldingerstraße
  - Dept. Urology, University Hospital Tübingen, Tübingen, Hoppe-Seyler-Straße 3

IPD SHARING:
Plan to Share IPD: No